CLINICAL TRIAL: NCT05334940
Title: Atopy Network - Comprehensive Allergy Centers: Medical Care of Patients With Moderate to Severe Allergic Diseases
Acronym: ATAC
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Margitta Worm, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: Atopy Registry
Record Dates: First submitted 2022-03-15; First posted 2022-04-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Atopic Disorders
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — optional blood sampling, stool sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic disorders: Patients with at least 2 atopic disorders who are eligible for systemic therapy with biologics
  Interventions: Other: not applicable, observational study

INTERVENTIONS:
Other: not applicable, observational study — Patients do not receive intervention

SUMMARY:
The Atopy Registry aims to assess data about atopic disorders and their medical care in a standardized form. With this, the comparative efficacy, tolerability and safety of systemic therapies for atopic disorders should be investigated. An optional additional module "Bioanalytic" shall provide insights into further connections regarding immunology, genetics and microbiome.

DETAILED DESCRIPTION:
The prevalence of atopic disorders increased in the western countries within the past decades. Atopic disorders are among others: food allergy, atopic dermatitis, allergic rhinitis, bronchial asthma, chronic spontaneous urticaria, eosinophilic esophagitis and chronic rhinosinusitis with nasal polyposis.

Seriously affected patients often have coexisting atopic disorders. In fact, 60-75% of the patients with a severe atopic dermatitis also suffer from an allergic rhinoconjunctivitis and 40-50% from bronchial asthma. This leads to a decreased quality of life (LG) especially in seriously affected patients.

The treatment of atopic disorders is not standardized yet. The Atopy Registry should promote the creation of a Germany-wide registry for different atopic disorders.Furthermore, the registry should characterize the medical care of patients with atopic disorders (patient satisfaction, therapy order, treatment success). This study serves as a longterm observation und is designed to compare different systemic therapies, since head-to-head studies regarding the efficacy are still missing. The analysis of biomaterial is involved to state possible correlations between endotype and phenotype.

ELIGIBILITY:
Inclusion Criteria:

* patients are at least 6 years old
* patients with a proven moderate to severe atopic disorder who are planned to receive a biologic systemic therapy
* at least one additional proven atopic disorder

Exclusion Criteria:

* <2 atopic disorders
* poor compliance
* pregnancy or breastfeeding

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a moderate to severe primary atopic disorder and at least one additional secondary underlying atopic disease
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Comorbidity Food Allergy | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Food Allergy: Food Allergy Quality of Life Questionnaire (FAQLQ) (type-dependent 23-30 items, score between 0 and 6; mean of scores, minimum = 0, maximum = 6; higher score = higher impact on quality of life)
Comorbidity Atopic Dermatitis | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Atopic Dermatitis: Atopic Dermatitis-Control-Test (ADCT) (6 items, score between 0 and 4; sum, minimum = 0, maximum = 24; higher score = higher severity)
Comorbidity Bronchial Asthma | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Bronchial Asthma: Asthma-Control-Test (ACT) (5 items, score between 0 and 5; sum, minimum = 0, maximum = 25; higher score = better disease control)
Comorbidity Chronic rhinosinusitis with nasal polyps | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Chronic rhinosinusitis with nasal polyps: 22 Items Sino-Nasal Outcome Test (SNOT22) (22 items, score between 0 and 5; sum, minimum = 0, maximum = 110; higher score = higher impact on quality of life)
Comorbidity Chronic Spontaneous Urticaria | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Chronic Spointaneous Urticaria: Urticaria Control Test (UCT) (4 items, score between 0 and 5; sum, minimum = 0, maximum = 20; higher score = better control)
Comorbidity Eosinophilic Esophagitis | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Eosinophilic Esophagitis: Dysphagia Symptoms Questionnaire (DSQ) (4 items, score between 0 and 4 but question-dependent; sum, minimum = 0, maximum = 10; higher score = higher impact)
Comorbidity Allergic Rhinitis | 3 years
  Improvement of at least one comorbidity with biologics therapy using a standardized questionnaire to assess disease severity for the following atopic diseases:
  Allergic Rhinitis: Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) (28 items, score between 0 and 6; mean, minimum = 0, maximum = 6; higher score = higher impact on quality of life)

SECONDARY OUTCOMES:
Food Allergy Severity | 3 years
  Altered assessment of severity by investigation of oral thresholds and accidental reactions by oral food challenge.
Atopic Dermatitis Severity | 3 years
  Altered assessment of severity and/or LQ using the Eczema Area and Severity Index (EASI).
  (Eczema Area and Severity; minimum = 0, maximum = 72; higher numbers = higher severity)
Allergic Rhinitis Severity | 3 years
  Altered assessment of severity using the Total Nasal Symptom Score (TNSS). (Total Nasal Symptom Score; 3 items, score between 0 and 3; minimum = 0, maximum = 9; higher score = higher severity)
Bronchial Asthma Severity FVC | 3 years
  Altered assessment of severity using the lung function parameter Forced Vital Capacity (FVC)
Bronchial Asthma Severity FEV1 | 3 years
  Altered assessment of severity using the lung function parameter Forced Expiratory Volume in 1 second (FEV1)
Bronchial Asthma Severity FEF25-75 | 3 years
  Altered assessment of severity using the lung function parameter Forced expiratory flow 25-75 (FEF25-75).
Chronic Spontaneous Urticaria LQ (CUQ2oL) | 3 years
  Altered assessment of LQ using the Chronic Urticaria Questionnaire for Quality of Life (CUQ2oL).
  (Chronic Urticaria Questionnaire for Quality of Life; 23 items, score between 0 and 4; the score is calculated in percentage, minimum = 0%, maximum = 100%; higher percentage = lower quality of life)
Chronic Spontaneous Urticaria Severity (AECT) | 3 years
  Altered assessment of severity using the Angioedema Control Test (AECT). (Angioedema Control Test; 4 items, score between 0 and 4; minimum = 0, maximum = 16; lower score = higher severity)
Chronic Spontaneous Urticaria Severity (UAS7) | 3 years
  Altered assessment of severity and/or LQ using the 7-Days Urticaria Activity Score (UAS7).
  (7-Days Urticaria Activity Score; 2 items on 7 days, score between 0 and 3; minimum = 0, maximum = 42; higher score = higher severity)
Eosinophilic Esophagitis Severity and/or LQ | 3 years
  Altered assessment of LQ using the Pediatric Quality of Life Inventory Eosinophilic Esophagitis (PedsQLEoE).
  (Pediatric Quality of Life Inventory Eosinophilic Esophagitis; 33 items, score between 0 and 4; scores are graded on an 0-100 scale in opposite order (0=100, 1=75, 2=50, 3=25, 4=0); minimum = 0, maximum = 100; higher mean score = higher quality of life
Chronic Rhinosinusitis with Nasal Polyposis Severity | 3 years
  Altered assessment of severity using the Nasal Polyp Score. (Nasal Polyp Score; 2 items, score between 0 and 4; minimum = 0, maximum = 8; higher score = higher severity)

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof., Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided